CLINICAL TRIAL: NCT05158322
Title: Effectiveness of the Staphylococcus Aureus Decolonization Circuit in Reducing Infection at the Surgical Site in Patients Scheduled for Primary Arthroplasty in the Lower Limb
Brief Title: Effectiveness of the Decolonization Circuit of S. Aureus, Reducing Infection in Primary Arthroplasty of the Lower Limb
Status: Active, not recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francisco Zamora Carmona, Enfermero Práctica Avanzada, Corporacion Parc Tauli
Other Study IDs: DESCO-2021
Record Dates: First submitted 2021-11-25; First posted 2021-12-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Nurse's Role; Surgical Site Infection; Patient Satisfaction
Keywords: Decolonization S. Aureus
MeSH Terms: conditions — Surgical Wound Infection; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lower limb joint replacement surgery is one of the most prevalent globally. In our center, more than 400 lower limb arthroplasties (LLA) are performed annually. Developing a Surgical Site Infection (SSI) after (LLA) increases morbidity, mortality and healthcare costs. Staphylococcus aureus is the main causative agent of SSI and especially in LLA. One third of the population is a nasal carrier of Staphylococcus aureus, being a risk factor for patients who have to undergo knee replacement or hip replacement. Several studies have confirmed that the detection of S. aureus carriers and their subsequent decolonization reduces SSI rates

DETAILED DESCRIPTION:
Implementation of a screening of all patients who have to undergo lower limb arthroplasty in our center, decolonization of patients with a positive screening result for S. aureus and subsequent follow-up.The circuit is established in the following phases:

1. Preoperative Nurse Visit:

   Oral and written information on the study and procedure is given, the informed consent will be signed, and the sample (nasal swab) is collected from all patients scheduled for lower limb arthroplasty surgery in our center. The sample is sent to microbiology.

   It will be recorded in the computerized medical history.
2. Control of results:

   If the sample has been run by rapid circuit at 24 hours or conventional at 4 days, the Consultation Nurse reviews the results of the screened patients.

   c. In case of negative screening, patients follow the usual clinical practice circuit.

   d. In case of positive screening, the patients are summoned the next day to Consultations to give and explain the decolonization treatment.
3. Indication of decolonization to S. aureus:

   The following treatment is prescribed and facilitated in the nurse's office and will be recorded in the history:
   * Intranasal mupirocin every 8h. for 5 days (in case of resistance, intranasal fusidic acid is given every 12 hours for 5 days). Treatment is always carried out 7 days before the day of admission for surgery.
   * Chlorhexidine gluconate (single-dose sachets) daily shower until the day of admission for the intervention.
4. Post-decolonization control S. aureus:

   The patient is asked about adherence to treatment and a nasal smear is performed in the Presurgical Unit. In the event that the Innervencion is before the end of the treatment. It is not deprogrammed, but the treatment will continue until it is completed. The control nasal smear, in these cases, will be collected at the first treatment in the nurse's office. The satisfa
5. The patients will be followed for 6 weeks, a period in which an infection is considered an acute surgical site, it will be recorded if the infection is due to S. aureus.
6. The circuit will be evaluated in relation to efficacy and impact (number of patients operated on, number of screening, number of S. aureus positives, number of decolonizations and if they have been effective, number of S. aureus infections after The proposed intervention and treatment will be compared with the infections of the same period of the year 2019.ction survey of the decolonization protocol (VAS 0-10) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Patients who are going to undergo knee or hip replacement surgery.
* Patients with a positive result in the first nasal smear to S. aureus, and follow the decolonization protocol.
* Patients who give their informed consent to participate in the study.

Exclusion Criteria:

* Patients scheduled for VPE less than 2 days after surgery.
* Patients unable to give their informed consent freely. Inadequate cognitive ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who are going to be operated
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate with a VAS scale (0-10) the satisfaction of the participant with the information on the decolonization process of S. aureus. | 6 weeks
  The participant is satisfied with the information received throughout the decolonization. to be assessed with the EVA scale (0 not at all satisfied / 10 very satisfied)

SECONDARY OUTCOMES:
The participant evaluates his social well-being on the VAS scale (0-10) based on the care received by professionals throughout the S. aureus decolonization process. The number of patients who scored 9 or 10 on the VAS scale will be assessed as satisfied. | 6 weeks
  Number of participants who perceive well-being with the VAS scale (0 very dissatisfied / 10 very satisfied) linked to the quality of care throughout the decolonization process.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Zamora-Carmona, Nurse, Principal Investigator — Corporació Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain